CLINICAL TRIAL: NCT00405873
Title: A Prospective, Open, Single-arm, Multicenter Phase II Clinical Trial to Evaluate the Tumour Response and Safety in Patients With Advanced Primary Hepatocellular Carcinoma Treated With AMT2003
Brief Title: Study to Evaluate Tumour Response in Cancer Patients With Advanced Hepatocellular Carcinoma (Liver Cancer) With AMT2003
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Auron Healthcare GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMT/P2GI/001 Part I; LC004AURON2005
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Primary hepatocellular carcinoma; Liver cancer; Tumour response; Quality of life
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

ARMS (1):
- AMT2003 (Experimental)
  Interventions: Drug: AMT2003

INTERVENTIONS:
Drug: AMT2003

SUMMARY:
The purpose of the study is to evaluate the efficacy and the safety of AMT2003 in cancer patients with advanced primary hepatocellular carcinoma

The primary endpoint is best overall response rate within 20 weeks after registration

DETAILED DESCRIPTION:
The study will include patients with advanced primary hepatocellular carcinoma refractory to standard therapy or for which no effective standard therapy exists.

The best overall response rate is the best response recorded from the start of treatment until disease progression / recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Cancer confirmed by histology or cytology
* At least one measurable lesion
* Advanced disease refractory to standard therapy or for which no standard therapy exists
* Life expectancy of at least 3 months

Exclusion Criteria:

* Known secondary neoplasia or central nervous system (CNS) metastases; acute or chronic leukemia, lymphoma or multiple myeloma
* Body weight below 45 kg
* Female patients who are pregnant or breast feeding or adults of reproductive potential not employing effective method of birth control
* Confirmed diagnosis of HIV
* Insulin dependent diabetes mellitus / abnormal glucose tolerance test (GTT) / latent diabetes mellitus type I or II
* Chemotherapy or radiotherapy less than 4 weeks prior to entry
* Surgery less than 2 weeks prior to entry (or not recovered from effects of surgery)
* Participation in a clinical trial less than 30 days prior to entry into study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Best overall tumour response according to RECIST; within 20 weeks after registration; confirmation 6 +/- weeks later | March 2010

SECONDARY OUTCOMES:
Progression Free Survival (PFS) time | March 2010
Overall Survival (OS) time | March 2010
Quality of Life (EORTC QLQ-C30) and Performance Status (Karnofsky Index) | March 2010
Safety and Tolerability | March 2010

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Blum, Prof. Dr. med. Dr. h. c., Principal Investigator — University Hospital Freiburg
Locations (2):
- Germany (2):
  - University Hospital Freiburg, Dept. of Internal Medicine II, Freiburg im Breisgau, Baaden-Wuerttemberg
  - Clinic SanaFontis, Freiburg im Breisgau

REFERENCES:
- See also: Now legally responsible for study — http://www.alpiniainstitute.com